CLINICAL TRIAL: NCT04538638
Title: Mesenteric SParIng Versus Central mesenterectomY in Ileocolic Resection for Terminal Ileitis in Crohn's Disease
Acronym: SPICY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Willem A. Bemelman, Full professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL61632.018.18
Record Dates: First submitted 2020-08-31; First posted 2020-09-04 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Ileocolic; Mesenteric Sparing; Extended Mesenterectomy
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: Patients with Crohn's disease will be randomised in a 1:1 ratio for mesenteric sparing versus central mesenterectomy when performing an ileocolic resection for Crohn's disease
Who Masked: Participant, Care Provider
Masking Description: There is no blinding to the treatment allocation for the treating surgeon. The treatment will be blinded for the treating gastroenterologist, the endoscopist and the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenteric Sparing ileocolic resection (Active Comparator): Standard procedure for CD, ileocolic resection without removal of the mesentery.
  Interventions: Procedure: Mesenteric sparing ileocolic resection
- Central mesenterectomy ileocolic resection (Active Comparator): Experimental procedure for CD: ileocolic resection in which the mesentery is taken up to the level of the ileocolic trunc.
  Interventions: Procedure: Central mesenterectomy ileocolic resection

INTERVENTIONS:
Procedure: Mesenteric sparing ileocolic resection — Mesentery left in situ
  Arms: Mesenteric Sparing ileocolic resection
Procedure: Central mesenterectomy ileocolic resection — Mesentery is taken up to the level of the ileocolic trunk
  Arms: Central mesenterectomy ileocolic resection

SUMMARY:
The aim of this multicenter randomised controlled trial is to analyse the six month endoscopic recurrence following a mesenteric sparing versus a central mesenterectomy performing an ileocolic resection for CD.

DETAILED DESCRIPTION:
There is emerging evidence to suggest that Crohn's disease (CD) may be a disease of the mesentery rather than just of the bowel alone. A more extensive central mesenterectomy (up to the level of the ileocolic artery), in order to remove an increased volume of affected mesentery to prevent postoperative CD, has been suggested to lead to beneficial results. It is hypothesised that patients who undergo a central mesenterectomy during an ileocolic resection compared to a mesenteric sparing ileocolic resection will have decreased recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. Ileocolic disease with an indication for ileocecal resection
2. Concurrent therapies with corticosteroids, 5-ASA drugs, thiopurines, MTX, antibiotics, and anti-TNF therapy are permitted.
3. All patients should have undergone a colonoscopy and MR enterography (or CT enterography if MR contraindicated) in last 3 months to assess extent of disease.
4. Ability to comply with protocol.
5. Competent and able to provide written informed consent.
6. Patient must have been discussed in the local MDT

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Inability to give informed consent.
2. patients less than 16 years of age.
3. Patients undergoing repeated ileocolic resection.
4. Clinically significant medical conditions within the six months before the operation : e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the patient.
5. History of cancer < 5 years which might influence patients prognosis
6. Emergent operation.
7. Pregnant or breast feeding.
8. Inability to follow up at 3, 6 and 12 months for postoperative assessment, imaging and endoscopy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
The post-operative endoscopic recurrence of Crohn's disease at six months following ileocolic resection | 6 months after surgery

SECONDARY OUTCOMES:
Postoperative morbidity | 30 days after surgery
  Number of patients with Postoperative morbidity
Clinical recurrence rate following ileocolic resection | 1 year after surgery
  Number of patients with Clinical recurrence rate following ileocolic resection
The need for restarting immunosuppressive medication within the first year postoperatively for endoscopic or clinical recurrence | 1 year after surgery
  .The need for restarting immunosuppressive medication within the first year postoperatively for endoscopic or clinical recurrence
The 5 year reoperation rate for recurrence of disease at the anastomotic site. | 5 years
  The 5 year reoperation rate for recurrence of disease at the anastomotic site.

CONTACTS AND LOCATIONS:
Overall Officials: Christianne J Buskens, Principal Investigator — Amsterdam UMC, location AMC; Willem A Bemelman, Principal Investigator — Amsterdam UMC, location AMC
Locations (1):
- Amsterdam UMC - Location AMC, Amsterdam, Meibergdreef 9, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Does de Willebois EML; SPICY study group. Mesenteric SParIng versus extensive mesentereCtomY in primary ileocolic resection for ileocaecal Crohn's disease (SPICY): study protocol for randomized controlled trial. BJS Open. 2022 Jan 6;6(1):zrab136. doi: 10.1093/bjsopen/zrab136. PMID 35171266
- [Derived] van der Does de Willebois EML, Bellato V, Duijvestein M, van der Bilt JDW, van Dongen K, Spinelli A, D'Haens GR, Mundt MW, Furfaro F, Danese S, Vignali A, Bemelman WA, Buskens CJ; SPICY collaborator group. Effect of mesenteric sparing or extended resection in primary ileocolic resection for Crohn's disease on postoperative endoscopic recurrence (SPICY): an international, randomised controlled trial. Lancet Gastroenterol Hepatol. 2024 Sep;9(9):793-801. doi: 10.1016/S2468-1253(24)00097-9. Epub 2024 Jul 15. PMID 39025100

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT04538638/SAP_000.pdf